CLINICAL TRIAL: NCT03383939
Title: Effects of Inhaled Alpha-1-anti-trypsin on Proteolytic Activity in BAL of Bronchiectasis Patients With Chronic Bronchial Expectoration
Brief Title: Inhaled A1AT in Adult Stable Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Bayer (Industry); Sociedad Española de Neumología y Cirugía Torácica (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AC(HG) 44/95
Record Dates: First submitted 2017-09-27; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Bronchiectasis Adult
Keywords: bronchiectasis; alpha1-antitrypsin; neutrophilic elastase
MeSH Terms: conditions — Bronchiectasis; alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Intervention Model Description: 2 parallel groups of patients with bronchictasis were investigated: 1 receiving inhaled prolastina and 1 receiving placebo (saline solution) all bronchiectasis patients were initially compared with 10 control patients with no bronchiectasis
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Experimental): 10 patients randomly allocated received nebulised alpha1-antitrypsin 250mg (diluted in 10ml injectable solution) once a day during 1 month.
  Intervention: nebulised alpha1-antitrypsin 250mg (diluted in 10ml injectable solution) once a day during 1 month
  Interventions: Drug: Group A
- group B (Placebo Comparator): 9 patients randomly allocated received 10ml 0.9%NaCl saline solution nebulised once daily during 1 month.
  intervention: 10ml 0.9% Sodium Chloride saline solution nebulised once daily during 1 month.
  Interventions: Drug: Group B
- Control (No Intervention): 10 patients without bronchiectasis were initially compared wiht bronchiectasis patients (group A + B) to define baseline levels of A1-AT and neutrophil elastase in BAL

INTERVENTIONS:
Drug: Group A — one nebulization with 250mg alpha-1-antitrypsine diluted in 10ml injectable solution once a day during 1 month. A CR-60 high flow compressor and Ventstream nebulizer were used for nebulization.
  Other Names: inhaled Prolastin (nebulized alpha1-antitrypsin)
  Arms: group A
Drug: Group B — 10ml of 0.9% NaCl saline solution nebulised once daily for 1 month. A CR-60 high flow compressor and Ventstream nebulizer were used for nebulization.
  Other Names: placebo
  Arms: group B

SUMMARY:
Aim: to investigate the influence of alpha1-antitrypsin (A1-AT) nebulization on levels of A1-AT in BAL and plasma in patients with stable bronchiectasis.

Method: single-blind placebo-controlled randomised clinical trial. 19 stable bronchiectasis patients with chronic bronchial infection and 10 control patients (without bronchiectasis) underwent a bronchoscopy in order to assess levels and inhibitory capacity of A1AT and neutrophilic elastase. Afterwards, the 19 bronchiectasis patients were randomly allocated to receive inhaled A1AT 250mg diluted in 10ml 0.9% saline solution once a day for a month (Group A, n: 10) or placebo (10ml 0.9% saline solution; group B, n: 9). A new BAL was performed in both groups (A and B) 24 hours after the end of treatment (1month) to re-analyze A1AT and NE.

DETAILED DESCRIPTION:
Effects of inhaled alpha-1-anti-trypsin in bronchiectasis patients with chronic bronchial infection.

Introduction: one of the main features of bronchiectasis is chronic and deregulated neutrophilic bronchial inflammation. Excessive neutrophilic elastase (NE) activity has been widely described as part of the characteristic imbalance between proteases and anti-proteolytic enzymes that characterizes airways inflammation and progressive lung damage in bronchiectasis.

Alpha-1-antitrypsin (A1AT) is a protease inhibitor involved in protecting lung tissue from enzymes of inflammatory cells, including neutrophilic elastase, and its concentration rises in case of acute and chronic inflammation. Its reduction or absence is associated with the development of a specific kind of emphysema in case of exposure to tobacco smoking.

Moreover it is likely that its levels could be reduced in bronchiectasis as a consequence of chronic bronchial infection and inflammatory deregulation.

Aims:

1. concentrations of total and free NE, NE inhibitory capacity and A1AT levels were investigated in broncho-alveolar lavage (BAL) of bronchiectasis patients with chronic airways infection in stable conditions in comparison with a control group (patients without bronchiectasis)
2. The effects of inhaled A1AT (Prolastin) on BAL concentration of total and free NE and A1AT and inhibitory capacity of NE were assessed after one month of treatment in patients with bronchiectasis and chronic bronchial infection (placebo controlled trial) Study design: simple blind placebo-controlled randomized clinical trial

Methods:

19 patients with stable non cystic fibrosis bronchiectasis and chronic bronchial infection and 10 patients without bronchiectasis (control group) underwent a bronchoscopy to perform BAL analysis.

The 19 bronchiectasis patients were randomly allocated to receive inhaled A1AT 250mg diluted in 10ml 0.9% saline solution once a day for a month (Group A, n: 10) or placebo (10ml 0.9% saline solution; group B, n: 9). A new BAL was performed in both groups (A and B) 24 hours after the end of treatment (1month) to re-analyze A1AT and NE.

Clinical, microbiological, biochemical, functional and radiological characteristics of bronchiectasis and potential side effects of treatment on both arms were also recorded before (baseline), at 7, 15, 30 days of treatment and at 1 and 2 months follow-up visits after the end of treatment. The trial was approved by Spanish Ministry of Health (Trial nº 95/256) and local Ethics Committee (AC(HG) 44/95) and all patients signed written consent.

ELIGIBILITY:
Inclusion Criteria:

* Stable clinical conditions (no use of systemic antibiotic or steroid treatment in the last month)
* diagnosis of bronchiectasis bt CT scan
* chronic purulent or mucopurulent expectoration (daily sputum expectoration in the last 6 months or more)

Exclusion Criteria:

* Cystic fibrosis
* interstitial lung disease as cause of bronchiectasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1996-06-01 (Actual); Primary Completion 1999-09-07 (Actual); Study Completion 1999-09-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline BAL levels of A1AT | 1 MONTH
  Changes from baseline in levels of A1AT in broncho-alveolar lavage at 1 month of treatment with inhaled A1AT

SECONDARY OUTCOMES:
Changes from baseline neutrophil elastase in BAL | 1 month
  Changes from baseline in levels of neutrophil elastase in broncho-alveolar lavage at 1 month of treatment with inhaled A1AT
Changes from baseline neutrophil elastase inhibitory capacity in BAL | 1 month
  Changes from baseline in levels of neutrophil elastase inhibitory capacity in broncho-alveolar lavage at 1 month of treatment with inhaled A1AT

CONTACTS AND LOCATIONS:
Overall Officials: Javier De Gracia, MD, PhD, Principal Investigator — Servei de Pneumologia, Vall D'Hebron Hospital